CLINICAL TRIAL: NCT03284151
Title: Robotic and Focused Stereotactic Radiation Treatment of Good Prognosis Prostatic Adenocarcinoma
Brief Title: Focused Stereotactic Radiation Treatment of Prostatic Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Francois Baclesse, Luxembourg (Other)
Responsible Party: Sponsor
Other Study IDs: CYM6 Prostate CFB2
Record Dates: First submitted 2017-09-07; First posted 2017-09-15 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; good prognosis; focused treatment; Cyberknife
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Cyberknife

SUMMARY:
Focused stereotactic radiation treatment of localized prostatic adenocarcinoma. in order to quantify the delay between the focused treatment and the salvage procedure.

DETAILED DESCRIPTION:
Focused stereotactic radiation treatment of localized prostatic adenocarcinoma. in order to quantify the delay between the focused treatment and the salvage procedure.

Second objectives : objectives: prostate-specific antigen (PSA) response, MRI response, toxicity (CTCAEv4), quality of life (International Prostate Symptom Score (IPSS) and The International Index of Erectile Function (IIEF5) scores).

Method At first: Multiparametric Magnetic resonance imaging (MRI) - 12 biopsies within the whole gland.

Placement under endorectal ultrasound control of 4 fiducials at least 2 cm spaced.

Treatment : CyberKnife radiation treatment delivering 36.25 Gy in 5 fractions, in 10 days. Tracking using the 4 fiducials. Critical organs: Rectal and bladder wall: V35<2cc. Bladder neck and urethra: V35<1cc.

Salvage treatments: in such a context, salvage surgery or salvage intensity modulation radiation therapy (IMRT) treatments can in theory remain valid and safe options.

ELIGIBILITY:
Inclusion Criteria:

* Prostatic adenocarcinoma of Capra score≤2 invading no more than two adjacent of the 12 prostatic zones. Lesions>3mm. Maximal urinary flow rate ≥ 10ml/s, mean flow rate ≥ 5ml/s, post micturation volume ≤80ml, IPSS score ≤15.

Exclusion Criteria:

* systemic disease, ulcerative hemorrhagic ulcer or Crohn diseases, bladder neck stenosis, urethral implants, transurethral prostatectomy (TURP), any recurrent prostatitis within the last 3 years.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prostatic adenocarcinoma Capra≤2
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-01; Primary Completion 2020-01 (Actual); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Delay between the initial diagnosis and date of salvage treatment | through study completion, up to 36 months
  Delay between the initial diagnosis and date of salvage treatment

SECONDARY OUTCOMES:
PSA evaluation | 3, 6, 12, 18, 24, 30, 36 months
  PSA dosage
Birads score evaluation | 12, 24, 36 months
  Multiparametric prostatic MRI
Acute and late toxicity | 3, 6, 12, 18, 24, 30, 36 months
  Acute and late toxicity using the CTCAEv4
IPSS evaluation | 12, 24, 36 months
  IPSS score
IIEF5 evaluation | 12, 24, 36 months
  IIEF5 score

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Nickers, MD, PhD, Study Chair — Centre Francois Baclesse; Michel Untereiner, MD, Study Director — Centre Francois Baclesse
Locations (1):
- Centre Francois Baclesse, Esch-sur-Alzette, Luxembourg